CLINICAL TRIAL: NCT00216008
Title: Phase II Pharmacogenomic Study of Neoadjuvant Pre-irradiation Docetaxel and Cisplatin, Followed by Neoadjuvant Concomitant Docetaxel, Cisplatin and Irradiation, Followed by Surgery (CD-CDR-S) in Adult Patients With Operable Adenocarcinomas of the Esophagus or Gastroesophageal Junction
Brief Title: Pharmacogenomic Study of Docetaxel and Cisplatin, Followed by Docetaxel, Cisplatin and Irradiation.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Closure
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13946; USFIRB#103493; IIT 14069
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2009-07

CONDITIONS: Esophageal Adenocarcinomas; Adenocarcinomas of the Gastroesophageal Junction
MeSH Terms: interventions — Docetaxel; Cisplatin; Radiation; Surgical Procedures, Operative

INTERVENTIONS:
Drug: docetaxel
Drug: cisplatin
Procedure: radiation
Procedure: surgery

SUMMARY:
The purpose of this research study is to find out the effectiveness of the experimental combination of Docetaxel, Cisplatin, and radiation therapy administered prior to the surgical removal of your esophageal cancer.

DETAILED DESCRIPTION:
This study seeks to determine the safety and efficacy (the latter based on pathologic response rate, three- and five-year survival rates) of a three-phase multi-modality approach to adenocarcinomas of the esophagus or gastroesophageal junction. This study also aims retrospectively to determine if a specific tumor gene array profile would predict for pathologic complete response. Study schema is as follows. Patients are first staged, next they receive induction Docetaxel and Cisplatin on days 1 and 22, patients are then restaged, next they will undergo radiation therapy combined with Cisplatin and Docetaxel for approximately days 42 thorough 84, patients are again restaged, and finally surgery at approximately days 100 to 150.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmed esophageal adenocarcinoma or adenocarcinoma of the gastroesophageal junction (this diagnosis will be rendered by the gastroenterology endoscopist, and refers to tumors at the junction of the esophagus and the stomach, where >50% of the tumor mass is above the diaphragm). Tumors must not have greater than 2cm extension into the the cardia.
* Stage T2N0M0, T3N0M0, T1-3N1M0, T1-3N0-1M1a as determined by imaging studies and endoscopic ultrasound staging. M1a disease (celiac nodal metastasis) is permitted if other eligibility criteria are met. Any lesion suspicious for metastasis should biopsied (either by tru cut or fine needle aspiration) to prove eligibility.
* The subject has been deemed an appropriate surgical candidate by one of the surgical subinvestigators (ie. Not T4).
* No medical comorbidity making the patient not a surgical candidate.
* Subject must be 18 years or older
* Subject must understand the consent and be willing to give written and informed consent to participate in this investigational protocol, and for a tumor biopsy to be performed for research purposes at the time of their staging endoscopic ultrasound (clinically required for their care), and for a portion of their resection specimen be subjected to experimental laboratory analysis
* ECOG performance status <1 (Karnofsky >80%; see Appendix A).
* Subjects must have adequate caloric intake, as determined by a nutrition evaluation by a registered dietician. Nutrition intake may be enteral, hyperalimentation by enteral feeding tube, or by parenteral nutrition.
* Patients must have normal organ and marrow function as defined as: leukocytes >3,000/mcL; absolute neutrophil count >1,500/mcL; platelets >100,000/mcL; hemoglobin > 8 g/dl; Creatinine clearance (estimated by Cockroft-Gault equation) >50-mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Hepatic: Total bilirubin must be < ULN; AST and ALT and alkaline phosphatase must both be less than 2.5 x ULN.
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential).

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Common Toxicity Criteria Adverse Events version 3 (CTCAEv3) greater than grade 1 peripheral neuropathy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Pregnant and nursing women are excluded from this study. Women / men of childbearing potential not using a reliable and appropriate contraceptive method. Woman of childbearing potential with either a positive or no pregnancy test at baseline. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration
* Patients with a history of severe hypersensitivity reaction to docetaxel, cisplatin, or drugs formulated with polysorbate (Tween) 80.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with cisplatin and docetaxel or other agents administered during the study.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* History of clinically significant interstitial lung disease and/or pulmonary fibrosis.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Clinical or radiographic evidence of a tracheobronchial fistula or invasion of the aorta (i.e. T4 disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
toxicity and tolerability of this induction strategy
time to progression
surgical complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Chris Garrett, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States